CLINICAL TRIAL: NCT04175769
Title: Exploring the Effects of a Nutritional Supplement During Immunotherapy or Combination of Immunotherapy and Chemotherapy in Non-small Cell Lung Cancer Patients
Brief Title: A Nutritional Supplement to Support People With Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIT-0001
Record Dates: First submitted 2018-07-09; First posted 2019-11-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): Standard intervention of immunotherapy or combination of immunotherapy and chemotherapy, plus the experimental intervention nutritional product.
  Interventions: Dietary Supplement: Nutritional supplement
- Non-experimental intervention (Placebo Comparator): Standard intervention of immunotherapy or combination of immunotherapy and chemotherapy, plus the non-experimental intervention placebo product.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional supplement — Subjects will orally consume two gelatin capsules of nutritional supplement (1 gram), 2 times per day with meals, and 1 capsule at one additional meal or snack, totaling five capsules per day beginning the first day of treatment and continuing for the duration of their treatment.
  Arms: Experimental intervention
Other: Placebo — Subjects will orally consume two gelatin capsules of placebo (1 gram), 2 times per day with meals, and 1 capsule at one additional meal or snack, totaling five capsules per day beginning the first day of treatment and continuing for the duration of their treatment.
  Arms: Non-experimental intervention

SUMMARY:
People with non-small cell lung cancer are at risk for nutritional deficiencies.

The purpose of this study is to find out what effects a nutritional product has on patient's response to immunotherapy or combination of immunotherapy and chemotherapy. To do this, some of the participants will get the nutritional product and some will receive a placebo (a substance that looks like the study drug but does not have any active or medicinal ingredients). A placebo is used to make the results of the study more reliable.

Participants will be randomized to any of the following treatment groups:

- Group 1 (Experimental intervention): standard intervention of immunotherapy or combination of immunotherapy and chemotherapy plus the experimental intervention nutritional product.

Group 2 (Non-experimental intervention): standard intervention of immunotherapy or combination of immunotherapy and chemotherapy plus the non-experimental intervention placebo product.

Participants will take 5 capsules each day by mouth, starting on the first day of immunotherapy with or without chemotherapy and stopping upon completion of their immunotherapy with or without chemotherapy treatment.

Participants will complete a diary of their nutritional/ placebo product intake and will undergo the following assessments:

* Physical examination.
* Height and weight.
* ECOG status (the physician will record the impact on the cancer on daily living abilities).
* Concomitant medications recording.
* Adverse Event Assessment
* Computed tomography (CT) scan. A series of x-rays of the body from many angles that are turned into 3-dimensional pictures on a screen.
* Quality of life questionnaires.
* Blood collection

ELIGIBILITY:
Subject inclusion criteria

1. Systemic therapy-naïve patients with a histologically confirmed diagnosis of incurable or metastatic stage IIIB/IV non-small cell lung cancer with no EGFR and ALK mutation, who have agreed to receive chemotherapy or both immunotherapy and chemotherapy. Patients who have received prior platinum-based chemotherapy +/- immunotherapy in the curative setting will be allowed to enroll as long as the curative therapy ended at least 12 months prior to enrolment.
2. Age > or = 18 years.
3. A diagnostic CT image taken with a maximum of 60 days before initiation of systemic therapy.
4. An Eastern Cooperative Oncology Group Performance Status of ≤ 2.
5. Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.

Subject exclusion criteria.

1. Prior other malignancy, active (i.e., requiring treatment or intervention) within the previous 2 years, except for locally curable malignancies that have been apparently cured, which are allowed, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
2. Life expectancy <6 months at the discretion of the treating physician
3. Patients currently taking a supplement containing the nutritional supplement under study. Patients should have stopped taking supplements containing the nutritional supplement under study at least 30 days prior to enrolment.
4. A known hypersensitivity / allergy to the investigational product, placebo or to any ingredient in their formulations (e.g. gelatin or glycerin).
5. Enrolment in any other clinical protocol or investigational study with an interventional agent or assessments that may interfere with study procedures.
6. Weight loss >10% over past 6 months (weight 6 months ago minus weight today, divided by weight 6 months ago) x 100 = weight loss%.
7. Blood transfusions within 2 weeks of blood collection for the trial.
8. Untreated brain metastases (patients with previously resected and/or radiated brain metastases without neurologic symptoms are permitted).
9. Subject requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to study drug administration. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone, 2 mg per day of dexamethasone or up to 10 mg per day of prednisone) are allowed. Patients may take corticosteroids for ≤4 days as part of routine cancer-directed therapy prophylaxis (e.g., chemotherapy-induced nausea and vomiting).
10. Active autoimmune disease. Subjects with type 1 diabetes mellitus, stable endocrinopathies maintained on appropriate replacement therapy and skin disorders (e.g., vitiligo, psoriasis or alopecia) not requiring systemic treatment are allowed.
11. Uncontrolled diabetes, i.e. with random blood glucose >15.0 mmol/L.
12. Current or expected difficulty or inability to swallow capsules.
13. Use of non-steroidal anti-inflammatory drugs (NSAIDs) for ≥7 consecutive days. Patients are allowed to receive single doses of NSAIDs and may take daily 81 mg ASA.
14. In the investigators' opinion, patients who have medical conditions that could interfere with drug metabolism or absorption (e.g., short bowel syndrome, history of small bowel obstruction, Crohn's disease, etc.)
15. Serum albumin <35 g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | Upon completion of 4 cycles of treatment (each cycle is 21-days)
  Disease control rate is defined as the sum of patients with a complete response, partial response or stable disease via RECIST v.1.1 or iRECIST after 4-cycles of immunotherapy or a combination of chemotherapy and immunotherapy.

SECONDARY OUTCOMES:
Progression-free survival | Analysis will occur once 1-year survival data has been collected for all study participants.
  Defined as the time from treatment to time of documented disease progression or death. The RECIST v 1.1 or iRECIST will be used as the standardized tumor response assessment on CT images to determine disease progression.
1-year survival | Analysis will occur once 1-year survival data has been collected for all study participants.
  1-year survival (or death before 1-year)
Systemic therapy-induced toxicities | On day 1 of each treatment cycle (each cycle is 21 days) and at the end of treatment visit (within 30 days of last dose)
  Toxicity will be assessed and graded using the National Cancer Institute CTCAE, version 5.0.
Change in skeletal muscle mass and adipose tissue | Upon completion of 4 cycles of chemotherapy (each cycle is 21 days)
  Changes in cross-sectional areas of skeletal muscle will determined using two consecutive CT images from the third lumbar vertebrae region and normalized for stature (cm²/m²).
Change in Serum CRP | Upon completion of 4 cycles of chemotherapy (each cycle is 21 days)
  Serum CRP will be determined using enzyme-linked immunosorbent assays.
Change in Serum Albumin | Upon completion of 4 cycles of chemotherapy (each cycle is 21 days)
  Serum albumin will be determined using enzyme-linked immunosorbent assays.
Change in Fatty Acid Incorporation and Omega-3 Index | On day 1 of each treatment cycle (each cycle is 21 days) and at the end of treatment visit (within 30 days of last dose)
  A phospholipid analysis will be performed on blood samples collected prior to treatment on day 1 of cycles 1-4 and the end of treatment visit. Omega 3-Index will be calculated from the results of the phospholipid analysis.
Changes in Quality of Life via PROMIS Global Health Scale | Questionnaire will be administered at cycle 1 day 1, cycle 3 day 1 (each cycle is 21 days) and at the end of treatment (within 30 days of last dose).
  The PROMIS Global Health Scale v1.2 will be administered at cycle 1, 3 and at the end of treatment visit. The questionnaire will be scored according to the scoring manual, and changes analyzed to asses the effect of the investigational product on quality of life during treatment.
Changes in Quality of Life via PROMIS Physical Function Short Form | Questionnaire will be administered at cycle 1 day 1, cycle 3 day 1 (each cycle is 21 days) and at the end of treatment (within 30 days of last dose).
  The PROMIS Physical Function form v2.0 will be administered at cycle 1, 3 and at the end of treatment visit. The questionnaire will be scored according to the scoring manual, and changes analyzed to asses the effect of the investigational product on quality of life during treatment.
Changes in Quality of Life via FAACT | Questionnaire will be administered at cycle 1 day 1, cycle 3 day 1 (each cycle is 21 days) and at the end of treatment (within 30 days of last dose).
  The Functional Assessment of Anorexia Cachexia (FAACT) form version 4 will be administered at cycle 1, 3 and at the end of treatment visit. The questionnaire will be scored according to the scoring manual, and changes analyzed to asses the effect of the investigational product on quality of life during treatment.
Changes in Quality of Life via Taste and Smell Survey | Questionnaire will be administered at cycle 1 day 1, cycle 3 day 1 (each cycle is 21 days) and at the end of treatment (within 30 days of last dose).
  The Taste and Smell Survey v29Oct2015 will be administered at cycle 1, 3 and at the end of treatment visit. The questionnaire will be scored according to the scoring manual, and changes analyzed to asses the effect of the investigational product on quality of life during treatment.
Disease Control Rate after 2 cycles | Upon completion of 2 cycles of treatment (each cycle is 21-days)
  Disease control rate is defined as the sum of patients with a complete response, partial response or stable disease after 2 cycles of systemic therapy divided by the number of patients in the group. The Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or iRECIST will be used as the standardized tumor response assessment on CT images.

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada